CLINICAL TRIAL: NCT07320417
Title: Schneider Membrane Preservation Combined With In Situ Osteogenesis Strategy: A Feasibility Study of a Modified Maxillary Resection
Brief Title: Schneider Membrane Preservation With In Situ Osteogenesis: A Modified Maxillary Resection Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhao Guan (Other)
Responsible Party: Sponsor-Investigator, Wenzhao Guan, Attending Physician, Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2025]YX No. 175
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Diseases
MeSH Terms: conditions — Maxillary Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Procedure Group (No Intervention)
- Modified Procedure Group (Active Comparator)
  Interventions: Procedure: chneiderian Membrane-Preserving

INTERVENTIONS:
Procedure: chneiderian Membrane-Preserving — 1. Perform preoperative imaging evaluation of the patient to observe the condition of the maxillary sinus bony walls. During surgery, flap the tissue to expose the anterior wall of the maxilla, and create a window in the normal bone area of the anterior wall (approximately 10×15mm in diameter); 5. Carefully insert the maxillary sinus elevation instrument between the maxillary sinus membrane and the maxilla, delicately separate the maxillary sinus membrane while maintaining its integrity, and elevate the membrane to the required height.
  6. Place a wet gauze between the elevated membrane and the maxilla to protect the Schneiderian membrane, use an ultrasonic osteotome or reciprocating saw to remove the pathological tissue, and confirm negative margins intraoperatively with frozen section.
  Arms: Modified Procedure Group

SUMMARY:
This case series study aimed to find out if a new surgical technique that preserves the sinus membrane during upper jaw removal can help patients regenerate bone and recover function better after surgery. The study included two female patients with jaw tumors who were not suitable for or did not want complex reconstruction with tissue flaps. The main questions the study tried to answer were:

Can the preserved sinus membrane help new bone grow spontaneously in the jaw defect area after surgery? Can this new method reduce common complications seen with traditional surgery, such as oronasal fistula and empty nose syndrome? How well can patients recover in terms of chewing, swallowing, speech, and quality of life after the procedure?

In the study, during surgery, the surgeon carefully separated and preserved the sinus membrane from the bone that needed to be removed. After surgery, patients were followed with regular CT scans to check new bone growth. They also underwent tests to measure chewing force, swallowing ability, speech function, and quality of life to evaluate the long-term outcomes of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary lesions requiring resection of the jaw as diagnosed by imaging (CT) and pathology;
* CT shows the lesion only invades the maxilla without involving the maxillary sinus cavity;
* No nasal septum within the maxillary sinus cavity, with an intact and smooth sinus floor bone wall;
* No distant metastatic malignant tumors;
* American Society of Anesthesiologists (ASA) classification I-III, able to tolerate general anesthesia.

Exclusion Criteria:

* Lesions invading the maxillary sinus mucosa;
* Presence of septa or severe inflammation in the maxillary sinus;
* Previous history of head and neck radiotherapy;
* Coexisting immune system diseases or metabolic bone diseases;
* Pregnancy or breastfeeding;
* Any surgical contraindications;
* Mental illness or inability to comply with follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Bone regeneration status | 6 months
  Patients were followed up at 1, 3, and 6 months to assess bone formation in the maxillary sinus floor (CT slices used the contralateral first maxillary molar in the surgical area as an anatomical reference for preoperative and postoperative comparison). Specifically, the Planmeca ProMax® 3D tool was used to evaluate bone regeneration, measuring the length in the coronal plane, the length in the sagittal plane, and the height (in mm) on CT scans. The volume of newly formed maxillary sinus floor bone (in cubic millimeters) was calculated to assess the newly generated bone in the maxillary sinus floor.

SECONDARY OUTCOMES:
Postoperative complications | 1 year
  One year after surgery, the patient underwent follow-up to detect the occurrence of complications such as oronasal fistula and empty nose syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shanxi Medical University, Shanxi, China